CLINICAL TRIAL: NCT00566579
Title: Cryotherapy for Human Papillomavirus Clearance in Biopsy-confirmed Cervical Low-grade Squamous Intraepithelial Lesions: a Randomized Controlled Trial
Brief Title: Cryotherapy for Human Papillomavirus Clearance in Biopsy-confirmed Cervical Low-grade Squamous Intraepithelial Lesions
Acronym: Cryotherapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of additional funding
Sponsor: Khon Kaen University (Other)
Responsible Party: Clinical Epidemiology Unit (CEU), Faculty of Medicine, Khon Kaen University, Thailand
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HE500830
Record Dates: First submitted 2007-11-30; First posted 2007-12-03 (Estimated); Results first posted 2010-08-02 (Estimated); Last update posted 2010-08-10 (Estimated); Status verified 2007-12

CONDITIONS: Human Papillomavirus Clearance at 12 Months
Keywords: Human papillomavirus; Clearance; Cryotherapy
MeSH Terms: interventions — Cryotherapy; Cryosurgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Double-freezing cryotherapy was done within one month after the primary hpv testing was positive. Pap smear and colposcopy were done at 6 months and 12 months. HPV testing was repeated again at 12 months.
  Interventions: Procedure: Cryotherapy
- B (No Intervention): Pap smear and colposcopy were done at 6 months and 12 months. HPV testing was repeated again at 12 months.

INTERVENTIONS:
Procedure: Cryotherapy — Double freezing technique
  Other Names: Cryosurgery
  Arms: A

SUMMARY:
Persistent human papillomavirus (HPV) infections is the single necessary cause of cervical cancer. Cervical cancer is still the major health problem in the developing countries. It has been the first rank women's cancer in Thailand for many decades. Approximately 10-20% of Thai women have the high-risk HPV (HR-HPV) infections in their cervices. This will frequently lead to low-grade squamous intraepithelial lesions (LSILs) (10%), high-grade squamous intraepithelial lesions (HSILs) (0.8%), and finally, cervical cancers (0.16%) within 10-20 years. The treatment options for LSILs are either observation or ablative surgery. However, in our institute, cryotherapy, which is the one of ablative surgery, is more frequently used to comfort our women. It is not only effective but safe with only minimal side effects; watery leukorrhea for 2-4 weeks, and local cervical infection not more than 1%. Contraindication to this procedure are active cervical infection, lesion of 2 mm-larger than probe, lesion inside cervical os and suspected cervical cancer. Additionally, in developing countries such as Thailand, this treatment is safe, acceptable, feasible and effective. Patients with LSILs could also have this treatment in some rural area from the 10-days trained nurses. Fortunately, recent reports showed that cryotherapy has abilities not only in clearing LSILs but also clearing the HPV infections, its necessary cause. However, there are no randomized controlled trial compared its clearing ability between observation and cryotherapy. Therefore, a randomized controlled trial is needed to demonstrate that. Findings from this trial will contribute enormously to older women who already get infected by HPV. Aside from preventing cervical cancer in treated woman, cryotherapy could also give her relief from worrying about having a time-bomb like HPV infection in her cervix.

DETAILED DESCRIPTION:
This will be a hospital-based, parallel, assessor-blinded, randomized controlled trial. Study subjects refer to LSIL patients, more than 30 years-old, with positive HPV testing who do not have any contraindication of performing cryotherapy. Therefore, after recruitment LSIL patients whose age more than 30 years-old, we will exclude only those who have negative HPV testing or any contraindications of performing cryotherapy. The primary outcome is HPV clearance (negative HPV testing for the baseline HPV type) at 12 months after the treatment. Subjects will be randomly allocated to be treated by cryotherapy or observation only by using block randomization with varied block size of 2, 4, and 6. The sample size of at least 25 for each arm was planned to have the power of 80% to detect 20% difference rates of HPV clearance after 12 months of treatment between the two arms, with significance level of 0.05, two-sided test.

Study population:

Biopsy-confirmed LSIL patients, age more than 30 years-old, referred to either Srinagarind Hospital's, Khon Kaen Hospital's, or Roi Et Hospital's colposcopic clinics.

Inclusion criteria:

* Baseline HPV testing is positive.
* Be able to give their informed consent to this study.

Exclusion criteria:

* Having active cervical infection
* Having lesion of 2 mm-larger than probe
* Having lesion inside cervical os
* Having suspected cervical cancer lesion

Sample and sample size:

From previous studies, HPV clearance rate after cryotherapy at 12 months is 83.9%. (Elfgren, 2002) Spontaneous HPV clearance rate in young women at 24 months is 70%. (Moscicki, 1998) However, this HPV clearance rate in women older than 34 years-old at 12 months is only 53.6%. (Clavel, 2005) Using these numbers respectively as PE and PC putting in the formula below, we can calculate our sample size in each group. The sample size will be calculated to detect the 20-40% difference between the HPV clearance rates after 12 months, at significant level of 95% and power of 80% (two-sided test), using the approach of Lachin that was reviewed in the paper of Donner.(Donner, 1984)

Required sample size at different rate of clearance

P-control P-experimental Alpha level Power N Difference 95%CI 0.50 0.70 5% 80% 103 20 6.9-33.1 0.50 0.75 5% 80% 66 25 9-41 0.50 0.80 5% 80% 45 30 11.3-48.7 0.50 0.85 5% 80% 33 35 14-56 0.50 0.90 5% 80% 25 40 17.1-62.9

The sample size of at least 25 patients in each group will be chosen because of its precision and feasibility. Such sample size can detect 40% difference of HPV clearance rate between the two groups, at 95% significant level, with the power of 80%, 95%CI of 17.1-62.9, respectively.

Instruments:

After signing on the consent form, all eligible patients will be examined by the baseline standard procedures and PCR-HPV testing for 37 HPV types. Only positive HPV testing ones will be enrolled in the trial and then randomized to receive the cryotherapy or observation. The method of block randomization, with block size varies from 2 to 6, will be used to allocate treatments.

The allocation ratio is 1:1. The allocation sequence will be generated by computer, using STATA software version 10.0.

Based on the obtained schedule, the number of sealed envelopes, which are equal to the required blocks, will be prepared and labeled. Each envelope contains the corresponding sealed allocation cards that will allocate treatments to patients.

Colposcopy and cryotherapy instruments are available in our colposcopic clinic. However, we will reimburse for all CO2-gases tanks and materials used for Pap smears and HPV testing.

The people, who prepare the randomized scheme, will not involve in the trial. The allocation schedule will be concealed to the assessor (who measure the HPV testing) until the end of trial.

Data collection and measurement:

Because of the difference between two treatments, only the assessor (who measure the HPV testing) will be blinded from the treatments.

The specimens will be sent to the assessor without patient's name or HN that can be linked to the treatment received. They will be provided only the study ID number in which only the principle investigator can link it to the treatment received.

The main outcome is HPV clearance. It is measured by the gold-standard HPV testing. This will be performed at baseline and 12 months later.

Data analysis:

There were two main parts of analysis - describing selected characteristics of the study patients and analysis for answering the research questions. The first part, selected baseline characteristics of the patients in each treatment were compared i.e. age, sex, sexual experiences, underlying diseases, etc. Comparability of the distribution of those selected characteristics based on judgment rather than statistical significant tests. In this part, proportion was use for summarizing categorical data. For continuous data, the statistics include mean, standard deviation, minimum, maximum, and median.

For the second part, the analysis was based on the group in which the study patients were randomized (intention-to-treat basis). The different rate of clearance between the two arms of the trial and its 95% confidence interval will be calculated. This will be done at 12 months after the treatment. Z-test will be used for testing if such differences are different from zero. Multiple logistic regression will be used to control effects of any important confounding factors. Absolute risk reduction (ARR), relative risk reduction (RRR) and number needed to treat (NNT) will also be calculated.

The statistical analysis of this clinical trial will be performed based on intention-to-treat principle. All hypothesis tests are two-tailed at significant level of 0.05. Statistical package for all analysis is STATA version 10.0.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-confirmed LSIL patients
* Age more than 30 years-old
* Baseline HPV testing is positive.
* Be able to give their informed consent to this study.

Exclusion Criteria:

* Having active cervical infection
* Having lesion of 2 mm-larger than probe
* Having lesion inside cervical os
* Having suspected cervical cancer lesion

Min Age: 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-12; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bandit Chumworathayi, MD, Principal Investigator — Gynecologic Oncology Division, OBGYN Department, Faculty of Medicine, Khon Kaen University
Locations (1):
- Srinagarind Hospital, Faculty of Medicine, Khon Kaen University, Muang, Changwat Khon Kaen, Thailand

REFERENCES:
- [Derived] Chumworathayi B, Thinkhamrop J, Blumenthal PD, Thinkhamrop B, Pientong C, Ekalaksananan T. Cryotherapy for HPV clearance in women with biopsy-confirmed cervical low-grade squamous intraepithelial lesions. Int J Gynaecol Obstet. 2010 Feb;108(2):119-22. doi: 10.1016/j.ijgo.2009.09.012. Epub 2009 Nov 4. PMID 19892345
- See also: The Thailand Research Fund's website — http://www.trf.or.th/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: During December 2007 to March 2009, 103 subjects who had been documented as LSIL from cervical biopsy histopathology were recruited from three colposcopic clinics.
Pre-assignment Details: 3 of them declined to participate in this study. Only 60 of these 100 cases had positive results for HPV testing. Among women who had positive HPV testing results, 29 were randomly allocated to receive cryotherapy and 31 were allocated to observation.
Groups:
- Cryotherapy: Double-freezing cryotherapy was done within one month after the primary hpv testing was positive. Pap smear and colposcopy were done at 6 months and 12 months. HPV testing was repeated again at 12 months.
- Observation: Pap smear and colposcopy were done at 6 months and 12 months. HPV testing was repeated again at 12 months.
Period: Overall Study
Arm/Group | Cryotherapy | Observation
Started | 29 | 31
Completed | 29 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cryotherapy | Observation | Total
Number analyzed (Participants) | 29 | 31 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 31 | 60
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 42.17 (7.86) | 40.71 (7.51) | 41.42 (7.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 31 | 60
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Thailand | 29 | 31 | 60

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Human Papillomavirus Clearance
Description: At 12 months after treatment, a patient with negative results for HPV testing of previous types was considered as a clearance.
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Cryotherapy | Observation
Number analyzed (Participants) | 29 | 31
participants | 26 | 28

ADVERSE EVENTS:
Arm/Group | Cryotherapy | Observation
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/31
Other Adverse Events (participants affected / at risk) | 1/29 | 2/31
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cryotherapy (N=29) | Observation (N=31)
HSIL (Reproductive system and breast disorders) | 1 (1) | 2 (2) — HSIL rates, found by LEEP after HSIL Pap smears in treated group and observed group, were both very low (3.4% vs. 6.5%, p=0.58 ).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No